CLINICAL TRIAL: NCT00002418
Title: A Phase II, 24-Week, Open-Label Study Designed to Evaluate the Pharmacokinetics, Safety, Tolerability, and Efficacy of Novel Combination Therapy With Videx (Didanosine), Zerit (Stavudine), Viramune (Nevirapine), and MKC-442 (With or Without Hydroxyurea) for the Treatment of HIV-1 Infection in Non-Nucleoside Reverse Transcriptase Inhibitor Naive Patients Who Failed Previous Protease Inhibitor Treatment
Brief Title: The Safety and Effectiveness of Didanosine Plus Stavudine Plus Nevirapine Combined With MKC-442 in HIV-Infected Patients Who Have Not Had Success With Protease Inhibitors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Boehringer Ingelheim (Industry); Triangle Pharmaceuticals (Industry)
Purpose: Treatment
Other Study IDs: 292D; ICC 601
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-08-14 (Estimated); Status verified 2000-03

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — emivirine; Hydroxyurea; Nevirapine; Stavudine; Didanosine

INTERVENTIONS:
Drug: Emivirine
Drug: Hydroxyurea
Drug: Nevirapine
Drug: Stavudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to see if it is safe and effective to give a new anti-HIV drug combination to HIV-infected patients who have never taken nonnucleoside reverse transcriptase inhibitors (NNRTIs) and who have failed to respond to protease inhibitors (PIs). The drug combination will contain didanosine (ddI) plus stavudine (d4T) plus nevirapine (NVP) plus MKC-442. Hydroxyurea (HU) may be added.

DETAILED DESCRIPTION:
Patients receive a regimen of didanosine, stavudine, nevirapine, and MKC-442 for 24 weeks. Throughout the study, patients are evaluated for changes from baseline in plasma HIV-1 RNA levels and lymphocyte subsets and for development of adverse events and toxicities. Patients who experience virologic failure have the option of adding hydroxyurea to their treatment regimen or discontinuing from the study. After Week 24, patients with documented virologic response may continue treatment with didanosine, stavudine, nevirapine, and MKC-442, and, if applicable, hydroxyurea until a change in virologic status occurs (i.e., the patient experiences virologic failure). Follow-up visits are conducted every 4 to 12 weeks until permanent discontinuation from the study.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are at least 18 years old.
* Are HIV-positive.
* Have experienced treatment failure on a previous anti-HIV drug combination that contained at least one protease inhibitor. Your viral load must be between 5,000 and 50,000 copies/ml after 6 months of continuous treatment with that drug combination.
* Agree to use a barrier method of birth control (such as condoms) during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have a history of certain serious medical conditions, including pancreatitis, neuropathy, untreated seizures, or AIDS-related cancers, except Kaposi's sarcoma (KS).
* Are enrolled in another anti-HIV drug study while participating in this study.
* Have ever taken NNRTIs (such as NVP or MKC-442).
* Have ever taken ddI or d4T.
* Have taken certain medications within 30 days prior to study entry, including medications that affect your immune system (such as corticosteroids, interleukin-2, or interferon).
* Abuse alcohol or drugs.
* Have received chemotherapy or radiation therapy within 30 days prior to study entry. (Local radiation therapy is allowed.)
* Are allergic to any of the study drugs.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Pacific Oaks Med Group, Beverly Hills, California
  - Univ of Colorado / Health Science Ctr, Denver, Colorado
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Brown Univ School of Medicine, Providence, Rhode Island
  - Hampton Roads Med Specialists, Hampton, Virginia